CLINICAL TRIAL: NCT00338065
Title: External Influences Upon Ocular Homeostasis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Karen Joos, Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Vanderbilt IRB# 010436
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Intraocular Pressure
Keywords: Intraocular Pressure
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Subjects with autonomic dysfunction (Experimental): Subjects with known autonomic dysfunction diagnoses as defined by the General Clinical Research Center (GCRC) such as pure autonomic failure, Postural orthostatic tachycardia syndrome (POTS), and Multiple System Atrophy( MSA).
  1. Intraocular pressures, blood pressures, and retinal thicknesses are measured with postural changes
  2. Intraocular pressures, blood pressures, and retinal thicknesses are measured with water drinking.
  Interventions: Behavioral: Postural change; Behavioral: Water drinking
- Primary open-angle glaucoma subjects (Experimental): Subjects diagnosed with primary open-angle glaucoma following a glaucoma specialist's examination.
  1. Intraocular pressures, blood pressures, and retinal thicknesses are measured with postural changes
  2. Intraocular pressures, blood pressures, and retinal thicknesses are measured with water drinking.
  Interventions: Behavioral: Postural change; Behavioral: Water drinking
- Subjects with normal-pressure glaucoma (Experimental): Subjects with open-angle glaucoma damage following a glaucoma specialist's examination without ever an intraocular pressure recording greater than 21 mm Hg.
  .1. Intraocular pressures, blood pressures, and retinal thicknesses are measured with postural changes
  2. Intraocular pressures, blood pressures, and retinal thicknesses are measured with water drinking.
  Interventions: Behavioral: Postural change; Behavioral: Water drinking
- Normal subjects (Active Comparator): Subjects without evidence of glaucoma or autonomic dysfunction.
  ..1. Intraocular pressures, blood pressures, and retinal thicknesses are measured with postural changes
  2. Intraocular pressures, blood pressures, and retinal thicknesses are measured with water drinking.
  Interventions: Behavioral: Postural change; Behavioral: Water drinking

INTERVENTIONS:
Behavioral: Postural change — Intraocular pressures, blood pressures, and retinal thicknesses are measured with postural changes
Behavioral: Water drinking — Intraocular pressures, blood pressures, and retinal thicknesses are measured with water drinking.

SUMMARY:
Our experiments are designed to test the overall hypothesis that position-dependent or water-dependent intra-ocular pressure (IOP) spikes occur in humans, and that these challenge ocular homeostasis.

DETAILED DESCRIPTION:
Glaucoma is the second leading cause of blindness in the United States, yet its pathogenesis is poorly understood. This is an insidious disorder since the loss of peripheral vision which occurs first usually is not noticed by the victim. Approximately 1 million people in the United States have glaucoma, but are not aware of it. Glaucoma is not always associated with elevated intraocular pressures so that vision screenings which measure just intraocular pressure without assessing the optic nerve will also miss these patients with glaucomatous damage. Therefore, patients are often diagnosed only when they have severe irreversible vision loss. Vascular insufficiency or abnormal autoregulation versus mechanical pressure damage has been proposed as a major factor in the development of glaucoma. Presently, therapy is based upon lowering intraocular pressure. If a contributing intermittent pressure elevation factor can be elucidated and characterized, specific treatment modalities may then be developed and their effectiveness can be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients with autonomic dysfunction
* Patients with open-angle glaucoma
* Patients with normal-pressure glaucoma
* Normal subjects

Exclusion criteria:

* Medical students
* Prisoners
* Pregnant women

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-06; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Intraocular Pressure | Within 1 day
  A change in intraocular pressure is measured after change in posture or drinking water.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Joos, MD,PhD, Principal Investigator — Vanderbilt Eye Institute
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Phillips L, Robertson D, Melson MR, Garland EM, Joos KM. Pediatric ptosis as a sign of treatable autonomic dysfunction. Am J Ophthalmol. 2013 Aug;156(2):370-374.e2. doi: 10.1016/j.ajo.2013.03.009. Epub 2013 Apr 24. PMID 23622564
- [Result] Shibao CA, Joos K, Phillips JA 3rd, Cogan J, Newman JH, Hamid R, Meiler J, Capra J, Sheehan J, Vetrini F, Yang Y, Black B, Diedrich A, Roberston D, Biaggioni I. Familial Autonomic Ganglionopathy Caused by Rare CHRNA3 Genetic Variants. Neurology. 2021 Jul 13;97(2):e145-e155. doi: 10.1212/WNL.0000000000012143. Epub 2021 May 4. PMID 33947782